CLINICAL TRIAL: NCT01402258
Title: Tailored Internet-administrated Treatment of Anxiety Symptoms for Young Adults
Brief Title: Internet-administrated Treatment of Anxiety Symptoms for Young Adults
Acronym: NOVA-IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA-FORSS-2011-150291
Record Dates: First submitted 2011-07-01; First posted 2011-07-26 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tailored Internet-delivered CBT (Experimental): Behavioral: Tailored Internet-delivered CBT
  Interventions: Behavioral: Tailored Internet-administrated CBT-Treatment

INTERVENTIONS:
Behavioral: Tailored Internet-administrated CBT-Treatment — This intervention contains 6-8 text-based self-help modules in which 4 modules are fixed (the first three and the last) and the rest are prescribed following the diagnostic telephone interview. These modules contain material on panic disorder, social phobia, stress management, assertiveness training, concentration, relaxation among other things.

SUMMARY:
The purpose of this study is to determine whether tailored internet-administrated CBT is a feasible approach in the treatment of anxiety symptoms and comorbid anxiety and depressive symptoms in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 16-25 years old
* Have anxiety symptoms and/or anxiety syndrome

Exclusion Criteria:

* Suicide prone
* Alcohol addiction
* Ongoing psychological treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety symptoms two weeks post treatment, at six months and at 12 months post treatment.

SECONDARY OUTCOMES:
Quality of Life Inventory (QOLI)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in quality of life statements two weeks post treatment, at six months and at 12 months post treatment.
Montgomery Åsberg Depression Rating Scale-Self Rated (MADRS-S)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in depressive symptoms two weeks post treatment, at six months and at 12 months post treatment.
Clinical Outcome in Routine Evaluation - Outcome Measure (CORE-OM)- Change from baseline | Two weeks pre treatment, two weeks post treatment, six months and 12 months post treatment
  Change from baseline in anxiety and depressive symptoms two weeks post treatment, at six months and at 12 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Department of Behavioral Sciences and Learning, Linköping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden